CLINICAL TRIAL: NCT07039032
Title: A Clinical Study on the Use of a Domestically Produced Three-dimensional Cardiac Electrophysiological Mapping System Combined With Pressure Monitoring Technology and Star Mapping Technology for the Treatment of Paroxysmal Atrial Fibrillation.
Acronym: paroxysmal at
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai MicroPort EP MedTech Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Gao Henggan, Gao henggan, Shanghai MicroPort EP MedTech Co., Ltd.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A.1
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Paroxysmal Atrial Fibrillation (PAF)
Keywords: PFA; PeAF; PFA/RF
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-centre, post-marketing study (Experimental): Validating the safety and efficacy of pressure monitoring technology and star-shaped marking technology for the treatment of paroxysmal atrial fibrillation
  Interventions: Device: FireMagic™ Magbot Ablation Catheter 、FireMagic™ TrueForce™ Ablation Catheter

INTERVENTIONS:
Device: FireMagic™ Magbot Ablation Catheter 、FireMagic™ TrueForce™ Ablation Catheter — 1. The pressure-sensing catheter primarily consists of electrodes, a catheter body, and a control handle. The catheter body comprises a high-torque body and a flexible tip, divided into an adjustable bending segment and a main segment. By pushing or pulling the handle at the proximal end of the catheter, the internal traction wire at the catheter tip can be activated to control the bending of the tip. The adjustable bending segment is fixed with four electrodes at regular intervals, including one tip electrode and three ring electrodes.
  2. The disposable star-shaped magnetoelectric positioning catheter is specifically designed for cardiac electrophysiological mapping. The distal end of the catheter has multiple 3F branches, each with multiple platinum-iridium electrodes for collecting cardiac electrophysiological signals. The distal end of the catheter features an adjustable bend design; pushing the button on the catheter forward will cause the distal end of the catheter to bend.

SUMMARY:
Validating the safety and efficacy of pressure monitoring technology and star-shaped marking technology for the treatment of paroxysmal atrial fibrillation

DETAILED DESCRIPTION:
This trial will select appropriate clinical cases at clinical centres, where authorised investigators will perform ablation surgery for paroxysmal atrial fibrillation using the trial product. Indicators such as immediate ablation success rate and treatment success rate within three months post-surgery will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age between 18 and 80 years old, male or non-pregnant female.
2. Confirmed diagnosis of paroxysmal atrial fibrillation requiring catheter radiofrequency ablation surgery.
3. Fully understands the treatment plan and voluntarily signs the informed consent form, willing to undergo the examinations, surgery, and follow-up required by the plan.

Exclusion Criteria:

1. Post-ablation for atrial fibrillation
2. Reproductive-age patients who cannot use effective contraception within 12 months of enrolment
3. Left atrial size ≥50 mm, left ventricular ejection fraction ≤40%
4. Left atrial thrombus
5. History of atrial septal defect repair or atrial myxoma
6. History of cerebrovascular disease within the past 3 months (including stroke or transient ischaemic attack)
7. History of cardiovascular events within the past 3 months (including acute myocardial infarction, coronary artery intervention or bypass surgery, artificial valve replacement or repair, or atrial or ventricular incision)
8. Patients with acute or severe systemic infection
9. Patients with severe liver or kidney disease
10. Patients with significant bleeding tendencies or haematological disorders
11. Patients with malignant tumours or end-stage diseases
12. Patients deemed ineligible for this trial by the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Three-month follow-up success rate after surgery | Postoperative 3-month
  Postoperative 3-month treatment success rate: Specifically refers to the proportion of participants who, during the 3-month follow-up period (after the washout period), did not experience any episodes of atrial fibrillation/atrial flutter/atrial tachycardia lasting ≥30 seconds, as confirmed by electrocardiogram (ECG), Holter monitoring, or equivalent rhythm monitoring methods (including single-lead ECG), without the use of Class I or Class III antiarrhythmic drugs, relative to the total number of enrolled participants.

SECONDARY OUTCOMES:
Immediate ablation success rate | On the day of the surgery
  This refers to the proportion of subjects who achieved electrical isolation after surgery among the total number of patients enrolled in the study. The verification method involves waiting for 20 minutes after successful pulmonary vein electrical isolation and then reconfirming pulmonary vein conduction block.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China